CLINICAL TRIAL: NCT04142710
Title: A Pragmatic Randomized Control Trial Comparing Telehealth With Standard Clinical Care in the Follow-up of Patients With Chronic Conditions Within the Primary Care Setting
Brief Title: Pragmatic Randomized Control Trial of Telehealth vs Standard Care in Follow-up of Patients With Chronic Conditions
Acronym: MAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo Economics (Unknown); Norwegian Centre for Rural Medicine (Unknown); Norsk Gallup Institutt AS (Unknown)
Responsible Party: Principal Investigator, Tor Iversen, Professor of Health Economics, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Medisinsk avstandsoppfølging
Record Dates: First submitted 2019-07-05; First posted 2019-10-29 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Chronic Disease; Diabetes; Vascular Diseases; Chronic Lung Disease; Cancer; Psychiatric Disorder
Keywords: telemedicine; telehealth; randomized control trial; chronic disease; health services research; primary health care; primary care nursing
MeSH Terms: conditions — Chronic Disease; Diabetes Mellitus; Vascular Diseases; Neoplasms; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Follow-up using telehealth solutions (Experimental): Participants in this arm are followed up using a telehealth solution, as specified by the National Directorate of Health at the local centre. The actual follow-up is personalized to the individual user. All users receive a tablet, which can be used to answer questions about own health and/or transmit clinical measurements.
  Interventions: Device: Telemedicine: tablet and possibly tools to perform measurements
- Standard clinical care (No Intervention): Participants in this arm receive standard clinical care in accordance with their medinal needs.
- Non-randomized follow-up using telehealth solutions (Experimental): Participants in this arm are followed up using a telehealth solution, as specified by the National Directorate of Health at the local centre. The actual follow-up is personalized to the individual user. All users receive a tablet, which can be used to answer questions about own health and/or transmit clinical measurements. This arm is not randomized, but otherwise identical to the randomized experimental arm.
  Interventions: Device: Telemedicine: tablet and possibly tools to perform measurements

INTERVENTIONS:
Device: Telemedicine: tablet and possibly tools to perform measurements — Users of telemedicine can answer simple questions about their health condition and/or perform measurements related to their health (e.g., blood pressure, blood sugar, oxygen saturation, weight) via a tablet or a similar device. The results are transferred from the measuring devices to the tablet so that users can easily see them and track their own results over time. The results are transmitted digitally to a follow-up service. The follow-up service contacts the patient in case of signs of deterioration or when measurements lie outside what is normal values for the individual. The follow-up service provides medical support and guidance based on the patient's needs and plan for follow-up, and will, in consultation with the patient, assess whether this should contact their GP/emergency room.
  Arms: Follow-up using telehealth solutions; Non-randomized follow-up using telehealth solutions

SUMMARY:
The Norwegian health authorities has initiated a three-year trial of telehealth solutions as part of the treatment of patients with chronic illness in the period 2018-2021. Within the trial, telehealth indicates that patients are followed-up outside health-care facilities using information and communication technologies (ICTs). Patients who are followed up using telehealth solutions can answer questions about their own health and/or perform measurements related to their health (e.g. blood pressure, blood glucose, oxygen measurement, weight) via a tablet according to a personalized schedule. The measurement values are transferred from the measuring devices to a tablet so that the users can easily see them and track their results over time. The results are also transmitted digitally to a follow-up service, a healthcare center with nurses, who contacts the patient when needed. The follow-up service provides medical support and guidance based on the patient's needs and planned follow-up, and will, in consultation with the user, evaluate whether the user should contact the general practitioner (GP) or emergency room.

The study population of the trial includes users with comprehensive medical needs, with medium to high risk of worsening of their condition, hospitalization or increased need for health and care services.

The evaluation includes three main parts: 1) An effect evaluation which is designed as a randomized control trial, 2) a cost-benefit analysis, and 3) a process evaluation which aims to provide recommendations for how to organize and implement telemedicine in clinical practice. The primary outcomes include physical and mental health state, patient experience and use of health services.

The effect evaluation is designed as a pragmatic open label multi-center randomized control trial, with two parallel arms with 300 patients in each arm. Patients are recruited between February 2019 and June 2020.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a considerable disease burden and comprehensive medical needs
* The patient has a chronic disease
* The patient has medium to high risk of worsening of their condition, hospitalization or increased need for health and care services
* The patient has a high consumption of healthcare services
* The patient has a reduced level of function
* The patient is motivated to use telehealth solutions
* The patient is likely to benefit from the use of telehealth solutions

Exclusion Criteria:

* The patient is not competent to consent
* The patient is unable to handle the tablet and the measuring equipment to be used
* The patient has a substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2019-02-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Mean change in health-related quality of life (EuroQol 5 Dimensions 5 Levels (EQ-5D-5L)) from baseline at 6 months | Measured as change from baseline to 6 months after inclusion
  Patient's assessment of her health-related quality of life using the EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) questionnaire. The scale goes from 0 to 1 where higher scores mean a better outcome.
Mean change in health-related quality of life (EuroQol 5 Dimensions 5 Levels (EQ-5D-5L)) from baseline at 12 months | Measured as change from baseline to 12 months after inclusion
  Patient's assessment of her health-related quality of life using the EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) questionnaire. The scale goes from 0 to 1 where higher scores mean a better outcome.
Mean change in health-related quality of life (EuroQol 5 Dimensions 5 Levels (EQ-5D-5L)) from baseline at 18 months | Measured as change from baseline to 18 months after inclusion
  Patient's assessment of her health-related quality of life using the EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) questionnaire. The scale goes from 0 to 1 where higher scores mean a better outcome.
Mean change in health-related quality of life (Visual Analogue Scale (VAS)) from baseline at 6 months | Measured as change from baseline to 6 months after inclusion
  Patient's assessment of her health-related quality of life using Visual Analogue Scale (VAS). The scale goes from 0 to 100 where higher scores mean a better outcome.
Mean change in health-related quality of life (Visual Analogue Scale (VAS)) from baseline at 12 months | Measured as change from baseline to 12 months after inclusion
  Patient's assessment of her health-related quality of life using Visual Analogue Scale (VAS). The scale goes from 0 to 100 where higher scores mean a better outcome.
Mean change in health-related quality of life (Visual Analogue Scale (VAS)) from baseline at 18 months | Measured as change from baseline to 18 months after inclusion
  Patient's assessment of her health-related quality of life using Visual Analogue Scale (VAS). The scale goes from 0 to 100 where higher scores mean a better outcome.
Mean change in overall satisfaction with treatment and follow-up from baseline at 6 months | Measured as change from baseline to 6 months after inclusion
  Patients are asked to assess their overall satisfaction with their health care services: "To what extent are you satisfied with the follow-up of your health?". Answers on a four point scale ranging from "Not satisfied at all" to "Very satisfied"
Mean change in overall satisfaction with treatment and follow-up from baseline at 12 months | Measured as change from baseline to 12 months after inclusion
  Patients are asked to assess their overall satisfaction with their health care services: "To what extent are you satisfied with the follow-up of your health?". Answers on a four point scale ranging from "Not satisfied at all" to "Very satisfied"
Mean change in overall satisfaction with treatment and follow-up from baseline at 18 months | Measured as change from baseline to 18 months after inclusion
  Patients are asked to assess their overall satisfaction with their health care services: "To what extent are you satisfied with the follow-up of your health?". Answers on a four point scale ranging from "Not satisfied at all" to "Very satisfied"
Change in yearly health and care cost per person from baseline at 12 months | Yearly health and care cost per person is calculated at baseline and at 12 months after inclusion.
  The total cost of health and care services per patient is calculated by combining information on the use of health and care services with information about private and public costs of health and care services. Yearly health and care cost per person at baseline is defined as the yearly cost 365 days before inclusion. Similarly, the health and care cost at 12 months in defined as the total cost in the first year after inclusion. The change in mean is the primary outcome measure. Other changes, such as distributional changes, may be of interest.

SECONDARY OUTCOMES:
Mean change in sleep quality from baseline at 6 months | Measured as change from baseline to 6 months after inclusion
  Participants are asked the following question: "If you think about the last 7 days, to what degree have you experienced the following a) had problems sleeping at night b) had problems sleeping too much?" Answers on a four point scale ranging from "Not at all" to "To a very large extent".
Mean change in sleep quality from baseline at 12 months | Measured as change from baseline to 12 months after inclusion
  Participants are asked the following question: "If you think about the last 7 days, to what degree have you experienced the following a) had problems sleeping at night b) had problems sleeping too much?" Answers on a four point scale ranging from "Not at all" to "To a very large extent".
Mean change in sleep quality from baseline at 18 months | Measured as change from baseline to 18 months after inclusion
  Participants are asked the following question: "If you think about the last 7 days, to what degree have you experienced the following a) had problems sleeping at night b) had problems sleeping too much?" Answers on a four point scale ranging from "Not at all" to "To a very large extent".
Mean change in patients' sense of control over their health situation from baseline at 6 months | Measured as change from baseline to 6 months after inclusion
  Participants are asked the following question: "To what extent do you feel that you have control over your health situation?" Answers on a four point scale ranging from "Not at all" to "To a very large extent".
Mean change in patients' sense of control over their health situation from baseline at 12 months | Measured as change from baseline to 12 months after inclusion
  Participants are asked the following question: "To what extent do you feel that you have control over your health situation?" Answers on a four point scale ranging from "Not at all" to "To a very large extent".
Mean change in patients' sense of control over their health situation from baseline at 18 months | Measured as change from baseline to 18 months after inclusion
  Participants are asked the following question: "To what extent do you feel that you have control over your health situation?" Answers on a four point scale ranging from "Not at all" to "To a very large extent".
Mean change in patients' satisfaction with involvement of the GP from baseline at 6 months | Measured as change from baseline to 6 months after inclusion
  Patients answer the question "To what extent do you experience your GP is sufficiently involved in the follow-up of your health?" Answers are reported on a four point scale: "Not at all" to "To a very large extent".
Mean change in patients' satisfaction with involvement of the GP from baseline at 12 months | Measured as change from baseline to 12 months after inclusion
  Patients answer the question "To what extent do you experience your GP is sufficiently involved in the follow-up of your health?" Answers are reported on a four point scale: "Not at all" to "To a very large extent".
Mean change in patients' satisfaction with involvement of the GP from baseline at 18 months | Measured as change from baseline to 18 months after inclusion
  Patients answer the question "To what extent do you experience your GP is sufficiently involved in the follow-up of your health?" Answers are reported on a four point scale: "Not at all" to "To a very large extent".
Mean change in patients' sense of user involvement from baseline at 6 months | Measured as change from baseline to 6 months after inclusion
  Patients are asked "To what extent do you experience that you have opportunity to contribute to your own treatment?" Answers are reported on a four point scale: "Not at all" to "To a very large extent".
Mean change in patients' sense of user involvement from baseline at 12 months | Measured as change from baseline to 12 months after inclusion
  Patients are asked "To what extent do you experience that you have opportunity to contribute to your own treatment?" Answers are reported on a four point scale: "Not at all" to "To a very large extent".
Mean change in patients' sense of user involvement from baseline at 18 months | Measured as change from baseline to 18 months after inclusion
  Patients are asked "To what extent do you experience that you have opportunity to contribute to your own treatment?" Answers are reported on a four point scale: "Not at all" to "To a very large extent".
Mean change in the patients' number of appointments with the GP services from baseline at 12 months | Yearly use of the GP services is calculated at baseline and at 12 months after inclusion.
  Yearly number of appointments with the GP services at baseline is defined as the yearly use 365 days before inclusion. Similarly, the yearly number of appointments with of the GP services at 12 months is defined as the use in the first year after inclusion. The mean change is the primary outcome measure.
Mean change in the patients' number of outpatient visits from baseline at 12 months | Yearly number of outpatient visits is calculated at baseline and at 12 months after inclusion.
  Yearly number of outpatient visits at baseline is defined as the yearly use 365 days before inclusion. Similarly, the yearly number of outpatient visits at 12 months is defined as the use in the first year after inclusion. The mean change is the primary outcome measure.
Mean change in the patients' number of inpatient visits from baseline at 12 months | Yearly number of inpatient visits is calculated at baseline and at 12 months after inclusion.
  Yearly number of inpatient visits at baseline is defined as the yearly cost 365 days before inclusion. Similarly, the yearly number of inpatient visits at 12 months is defined as the use in the first year after inclusion. The mean change is the primary outcome measure.
Mean change in the patients' duration of inpatient visits from baseline at 12 months | Total duration of inpatient visits is calculated at baseline and at 12 months after inclusion.
  Total duration of inpatient visits at baseline is defined as the total duration of inpatient visits 365 days before inclusion. Similarly, the total duration of inpatient visits at 12 months is defined as the total duration in the first year after inclusion. The mean change is the primary outcome measure.
Mean change in the patients' number of emergency room visits from baseline at 12 months | Yearly number of emergency room visits is calculated at baseline and at 12 months after inclusion.
  Yearly number of emergency room visits at baseline is defined as the yearly use 365 days before inclusion. Similarly, the yearly number of emergency room visits at 12 months is defined as the yearly use in the first year after inclusion. The mean change is the primary outcome measure.
Mean change in the patients' number of home nursing visits from baseline at 6 months | Use of home nursing visits is measured one month prior to inclusion and 6 months after inclusion.
  Use of home nursing visits before inclusion is measured as the total number of home nursing visits 30 to 60 days prior to inclusion. Use at 6 months is measured as the total number of home nursing visits 150 to 180 days after inclusion.
Mean change in the patients' number of home nursing visits from baseline at 12 months | Use of home nursing visits is measured one month prior to inclusion and 12 months after inclusion.
  Use of home nursing visits before inclusion is measured as the total number of home nursing visits 30 to 60 days prior to inclusion. Use at 12 months is measured as the total number of home nursing visits 335 to 365 days after inclusion.
Mean change in the patients' number of home nursing visits from baseline at 18 months | Use of home nursing visits is measured one month prior to inclusion and 18 months after inclusion.
  Use of home nursing visits before inclusion is measured as the total number of home nursing visits 30 to 60 days prior to inclusion. Use at 18 months is measured as the total number of home nursing visits 515 to 545 days after inclusion.
Mean change in the patients' duration of home nursing visits from baseline at 6 months | Total duration of home nursing visits is measured one month prior to inclusion and 6 months after inclusion.
  Total duration of home nursing visits before inclusion is measured as the total duration of home nursing visits 30 to 60 days prior to inclusion. Total duration at 6 months is measured as the total duration of home nursing visits 150 to 180 days after inclusion.
Mean change in the patients' duration of home nursing visits from baseline at 12 months | Total duration of home nursing visits is measured one month prior to inclusion and 12 months after inclusion.
  Total duration of home nursing visits before inclusion is measured as the total duration of home nursing visits 30 to 60 days prior to inclusion. Total duration at 12 months is measured as the total duration of home nursing visits 335 to 365 days after inclusion.
Mean change in the patients' duration of home nursing visits from baseline at 18 months | Total duration of home nursing visits is measured one month prior to inclusion and 18 months after inclusion.
  Total duration of home nursing visits before inclusion is measured as the total duration of home nursing visits 30 to 60 days prior to inclusion. Total duration at 18 months is measured as the total duration of home nursing visits 515 to 545 days after inclusion.
Mean change in the patients' number of municipal emergency day care unit visits from baseline at 6 months | Use of municipal emergency day care unit visits is measured one month prior to inclusion and 6 months after inclusion.
  Use of municipal emergency day care unit visits before inclusion is measured as the total number of municipal emergency day care unit visits 30 to 60 days prior to inclusion. Use at 6 months is measured as the total number of municipal emergency day care unit visits 150 to 180 days after inclusion.
Mean change in the patients' number of municipal emergency day care unit visits from baseline at 12 months | Use of municipal emergency day care unit visits is measured one month prior to inclusion and 12 months after inclusion.
  Use of municipal emergency day care unit visits before inclusion is measured as the total number of municipal emergency day care unit visits 30 to 60 days prior to inclusion. Use at 12 months is measured as the total number of municipal emergency day care unit visits 335 to 365 days after inclusion.
Mean change in the patients' number of municipal emergency day care unit visits from baseline at 18 months | Use of municipal emergency day care unit visits is measured one month prior to inclusion and 18 months after inclusion.
  Use of municipal emergency day care unit visits before inclusion is measured as the total number of municipal emergency day care unit visits 30 to 60 days prior to inclusion. Use at 18 months is measured as the total number of municipal emergency day care unit visits 515 to 545 days after inclusion.
Mean change in the patients' duration of municipal emergency day care unit visits from baseline at 6 months | Total duration of municipal emergency day care unit visits is measured one month prior to inclusion and 6 months after inclusion.
  Total duration of municipal emergency day care unit visits before inclusion is measured as the total duration of municipal emergency day care unit visits 30 to 60 days prior to inclusion. Total duration at 6 months is measured as the total duration of municipal emergency day care unit visits 150 to 180 days after inclusion.
Mean change in the patients' duration of municipal emergency day care unit visits from baseline at 12 months | Total duration of municipal emergency day care unit visits is measured one month prior to inclusion and 12 months after inclusion.
  Total duration of municipal emergency day care unit visits before inclusion is measured as the total duration of municipal emergency day care unit visits 30 to 60 days prior to inclusion. Total duration at 12 months is measured as the total duration of municipal emergency day care unit visits 335 to 365 days after inclusion.
Mean change in the patients' duration of municipal emergency day care unit visits from baseline at 18 months | Total duration of municipal emergency day care unit visits is measured one month prior to inclusion and 18 months after inclusion.
  Total duration of municipal emergency day care unit visits before inclusion is measured as the total duration of municipal emergency day care unit visits 30 to 60 days prior to inclusion. Total duration at 18 months is measured as the total duration of municipal emergency day care unit visits 515 to 545 days after inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Tor Iversen, Professor, Principal Investigator — University of Oslo
Locations (9):
- Norway (9):
  - Bodø municipality, Bodø
  - Eid municipality, Eidfjord
  - Ullensaker municipality, Jessheim
  - Kristiansand municipality, Kristiansand
  - Larvik municipality, Larvik
  - Gamle Oslo district, Oslo, Oslo
  - Grünerløkka district, Oslo, Oslo
  - Sagene ditrict, Oslo, Oslo
  - St.Hanshaugen district, Oslo, Oslo

IPD SHARING:
Plan to Share IPD: No
Researchers are not allowed to share individual patient data with other researchers.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT04142710/Prot_SAP_001.pdf
  • Informed Consent Form (2019-02-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT04142710/ICF_000.pdf